CLINICAL TRIAL: NCT05713604
Title: Validation of a New Clinical Questionnaire for the Evaluation of the Pathophysiological Mechanisms of Chronic Pain "MecPain".
Brief Title: "MecPain", a New Questionnaire to Assess Chronic Pain Mechanisms.
Acronym: MecPain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: Grenoble University Hospital
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain
Keywords: Neuropathic pain; Nociplastic pain; Nociceptive pain; Chronic pain mechanisms
MeSH Terms: conditions — Chronic Pain; Neuralgia; Nociplastic Pain; Nociceptive Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Validation of a new clinical questionnaire, called 'MecPain', including 12 questions, aimed at better defining the pathophysiological mechanisms of a chronic pain condition. This questionnaire includes 8 components/sub-components, reflecting various aspects of the 3 main mechanisms of chronic pain: nociceptive, neuropathic, nociplastic. A series of 240 patients with well-characterized chronic pain syndrome (for more than 6 months) of the nociceptive, neuropathic or nociplastic type will be recruited (80 patients per type of pain). The patients will be interviewed by a pain specialist to complete the 12 questions of the questionnaire during a routine visit in a Pain Center (CHU Grenobles Alpes, Grenoble, France or CHU Henri Mondor, Creteil, France). The scoring obtained with the 'MecPain' questionnaire will be compared to the presence of neuropathic pain assessed by two previously validated questionnaires, the 'DN4' and the 'PainDETECT' questionnaires. The expected outcome is a validation of the 'MecPain' questionnaire to provide a better understanding of the pathophysiological mechanisms relating to the presence of a chronic pain syndrome in a given patient.

DETAILED DESCRIPTION:
The main objective of this study is to specify the physiopathological mechanisms of a chronic pain syndrome according to 5 main components (+ 3 "sensory" sub-components) reflecting various aspects of the 3 main mechanisms of chronic pain: nociceptive, neuropathic, nociplastic.

A score will be assigned based on the answers to each of the 12 questions of the 'MecPain' questionnaire for each of the 8 components/sub-components mentioned above.

240 chronic pain patients will be included (in two centers), according to 3 categories: 80 patients with nociceptive pain (mechanical or inflammatory joint or spinal pain), 80 patients with neuropathic pain (painful peripheral neuropathy, neuralgia or radiculalgia, pain related with spinal cord or brain injury), and 80 patients with nociplastic pain (fibromyalgia, glossodynia, temporomandibular joint pain, irritable bowel syndrome, painful bladder syndrome).

ELIGIBILITY:
Inclusion Criteria:

* Presence of a chronic pain syndrome (pain for more than 6 months);
* well-characterized pain syndrome of the nociceptive, neuropathic or nociplastic type

Exclusion Criteria:

* Opposition to the use of data obtained in the context of standard clinical follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pain for more than 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2023-02-02 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
The scores of the various components of the 'MecPain' questionnaire | Six months
  A score will be assigned based on the answers to each of the 12 questions of the 'MecPain' questionnaire

SECONDARY OUTCOMES:
The scores of the'DN4' and 'PainDETECT' questionnaires | Six months
  Scores of the'DN4" ranging from 0 to 10 and scores 'PainDETECT' ranging from 0 to 38

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de GRENOBLE ALPES, Grenoble, Alpes
  - Henri Mondor, Paris

IPD SHARING:
Plan to Share IPD: No